CLINICAL TRIAL: NCT01282684
Title: A Phase 1 First in Human Double-Blind, Placebo-Controlled, Randomized, Single Ascending Dose Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of PLX5622 in Healthy Adult Volunteers
Brief Title: Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of PLX5622 in Healthy Adult Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Plexxikon (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PLX115-01
Record Dates: First submitted 2011-01-18; First posted 2011-01-25 (Estimated); Last update posted 2015-03-30 (Estimated); Status verified 2015-03

CONDITIONS: Healthy
Keywords: Safety; Tolerability; Pharmacokinetics; PLX5622
MeSH Terms: interventions — PLX5622

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (7):
- single oral dose of 200 mg PLX5622 (Active Comparator): 6 subjects will be randomized to take a single oral dose of PLX5622 and 2 subjects will be randomized to take placebo.
  Interventions: Drug: PLX5622
- single oral dose of 400 mg PLX5622 (Active Comparator): 6 subjects will be randomized to take a single oral dose of PLX5622 and 2 subjects will be randomized to take placebo.
  Interventions: Drug: PLX5622
- single oral dose of 800 mg PLX5622 (Active Comparator): 6 subjects will be randomized to take a single oral dose of PLX5622 and 2 subjects will be randomized to take placebo.
  Interventions: Drug: PLX5622
- single oral dose of 1600 mg PLX5622 (Active Comparator): 6 subjects will be randomized to take a single oral dose of PLX5622 and 2 subjects will be randomized to take placebo.
  Interventions: Drug: PLX5622
- single oral dose of 1000 mg PLX5622 (Active Comparator): 6 subjects will be randomized to take a single oral dose of PLX5622 and 2 subjects will be randomized to take placebo.
  Interventions: Drug: PLX5622
- single oral dose of 1400 mg PLX5622 (Active Comparator): 6 subjects will be randomized to take a single oral dose of PLX5622 and 2 subjects will be randomized to take placebo.
  Interventions: Drug: PLX5622
- Placebo (Placebo Comparator): 2 patients per cohort will be randomly assigned to take placebo. 12 patients total will be randomized to take placebo in this study.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: PLX5622 — PLX5622 drug substance is an achiral,small molecule Fms kinase inhibitor. The drug product is available in capsule form, to be taken orally, in dosage strengths of 25 mg and 100 mg with matching placebo
  Arms: single oral dose of 1000 mg PLX5622; single oral dose of 1400 mg PLX5622; single oral dose of 1600 mg PLX5622; single oral dose of 200 mg PLX5622; single oral dose of 400 mg PLX5622; single oral dose of 800 mg PLX5622
Drug: Placebo — Matching placebo for PLX5622.
  Arms: Placebo

SUMMARY:
The purpose of this study is to study the safety and tolerability of a single dose of PLX5622 in healthy, adult human volunteers. This will be the first time PLX5622 has been taken by humans.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult male and female subjects, 18-65 years of age inclusive
* BMI 18 to 32 kg/m2 inclusive
* Female subjects must be surgically sterile or postmenopausal for the past year and have a negative urine pregnancy test. Male subjects and their partners of childbearing potential must be willing to use two methods of contraception, one of which must be a barrier method (e.g. condom) for up to 90 days after the last study drug administration.
* Willing and able to remain in the clinical research unit as required by the protocol
* Willing and able to provide written informed consent prior to any study related procedures and to comply with all study requirements

Exclusion Criteria:

* History or presence of significant cardiovascular, pulmonary, hepatic, renal, hematologic, gastrointestinal, endocrine, immunologic, dermatologic, neurologic, or psychiatric disease
* History or presence of any disease, medical condition, or surgery, which may have an effect on drug absorption, metabolism, distribution, or excretion of the investigational product
* Laboratory test results (including hepatic and renal panels, complete blood count, chemistry panel, and urinalysis) that the investigator believes show clinically relevant significant abnormalities for the normal reference range
* Any abnormality in the ECG (including QTc ≥450 msec) that in the opinion of the investigator increases the risk of participating in the study
* History or presence of alcoholism or drug abuse within the year prior to dosing
* Tobacco use, either current or within 3 months prior to dosing
* Use of any prescription medications or herbal remedies within 14 days prior to dosing, or use of over-the-counter medications or vitamins within 7 days prior to dosing, unless approved by the Sponsor
* Donation of whole blood within 56 days prior to the study
* Plasma donation within 7 days prior to the study
* Participation in an investigational device study or receipt of an investigational drug within 4 weeks prior to dosing
* Positive urine test for drugs of abuse
* Confirmed HIV, hepatitis B, or hepatitis C infection

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2011-01; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
Safety-Number of patients with adverse events | 7 days
  Subjects will take one oral dose of PLX5622 on Day 1. Physical examinations, vital signs, 12-lead electrocardiograms (ECG), adverse events, hematology, serum chemistry, coagulation, and urinalysis will be used to assess safety throughout the Days 1-4 of the study and on the follow up study visit on day 7. Adverse events will be monitored and reviewed for safety issues/abnormal changes in the above mentioned tests.
Tolerability-Number of patients with adverse events | 7 days
  Subjects will take one oral dose of PLX5622 on Day 1. Physical examinations, vital signs, 12-lead electrocardiograms (ECG), adverse events, hematology, serum chemistry, coagulation, and urinalysis will be used to assess safety throughout the Days 1-4 of the study and on the follow up study visit on day 7. Adverse events will be monitored and reviewed for tolerability issues/abnormal changes in the above mentioned tests.

SECONDARY OUTCOMES:
Pharmacokinetic profile: Measurement of area under the plasma-concentration-time curve | 7 days
  Pharmacokinetic (PK) samples will be collected prior to dosing and at 0.5, 1, 2, 4, 8, 12, 24, 26, 48, 60 and 72 hours following dosing. The pharmacokinetic profile of plasma PLX5622 will be analyzed by measurement of area under the plasma concentration-time curve [AUC0-t, AUC0-inf, AUC0-24].
Pharmacokinetic evaulation: Measurement of Peak Concentration | 7 days
  Pharmacokinetic (PK) samples will be collected prior to dosing and at 0.5, 1, 2, 4, 8, 12, 24, 26, 48, 60 and 72 hours following dosing. The pharmacokinetic profile of plasma PLX5622 will be analyzed by measurement of peak concentration (Cmax) and time to peak concentration (Tmax).
Pharmacokinetic profile: Measurement of half life and terminal elimination rate constant | 7 Days
  Pharmacokinetic (PK) samples will be collected prior to dosing and at 0.5, 1, 2, 4, 8, 12, 24, 26, 48, 60 and 72 hours following dosing. The pharmacokinetic profile of plasma PLX5622 will be analyzed by measurement of half-life (T1/2), and terminal elimination rate constant (Kel).

CONTACTS AND LOCATIONS:
Overall Officials: Gregory Haugen, MD, Principal Investigator — Cetero Research, San Antonio
Locations (1):
- Cetero Research, Fargo, North Dakota, United States